CLINICAL TRIAL: NCT01040286
Title: The Efficacy and Safety of Flurbiprofen Chip Versus Chlorhexidine Chip (Periochip®) in Therapy of Adult Chronic Periodontitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dexcel Pharma Technologies Ltd. (Industry)
Responsible Party: Avi Avramoff, V.P R&D, Dexcel Pharma Technologies Ltd.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLI/012F
Record Dates: First submitted 2009-12-27; First posted 2009-12-29 (Estimated); Last update posted 2010-07-07 (Estimated); Status verified 2010-07

CONDITIONS: Periodontitis
Keywords: Subjects, age>21, with Chronic periodontal disease on natural teeth characterized by the presence of at least 2 teeth with periodontal; pockets of 5-9 mm in depth demonstrating bleeding on probing without involving the; apex of the tooth and confirmed by dental X-ray.
MeSH Terms: conditions — Periodontitis | interventions — Flurbiprofen; Chlorhexidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Flurbiprofen Chip (Experimental)
  Interventions: Drug: Flurbiprofen
- Chlorhexidine chip (Active Comparator)
  Interventions: Drug: Chlorhexidine

INTERVENTIONS:
Drug: Flurbiprofen — 2.0 mg
  Arms: Flurbiprofen Chip
Drug: Chlorhexidine — 2.5mg
  Arms: Chlorhexidine chip

SUMMARY:
The purpose of the study is to assess efficacy and safety of Flurbiprofen Chip versus Chlorhexidine chip (Periochip®) in therapy of adult chronic periodontitis.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent form
2. Good general health
3. Male or female subjects aged >21 years old
4. Availability for the 9 week duration of the study
5. Chronic periodontal disease on natural teeth characterized by the presence of at least 2 teeth with periodontal pockets of 5-9 mm in depth (potential target teeth) demonstrating bleeding on probing without involving the apex of the tooth and confirmed by dental X-ray.
6. Females of childbearing potential must be non-pregnant and non-lactating at entry and agree to use an adequate method (Oral or parenteral hormonal contraceptive; Intrauterine device; barrier and spermicide) of birth control during the study.

Exclusion Criteria:

1. An existing aggressive periodontitis.
2. Presence of oral local mechanical factors that could (in the opinion of the investigator) influence the outcome of the study.
3. Presence of orthodontic appliances, or any removable appliances, that impinge on the tissues being assessed.
4. Soft or hard tissue tumours of the oral cavity.
5. Presence of dental implant adjacent to target tooth.
6. Presence of more than 2 adjacent periodontal pockets on the same potential target tooth.
7. Periodontal pockets of more than 9 mm in depth, and/or with class 2 or 3 furcation involvement, on the potential target tooth.
8. Systemic antibiotic therapy or periodontal/mechanical/local delivery therapy within 6 weeks prior to study entry and throughout the study duration.
9. History of allergy to chlorhexidine, flurbiprofen or to other non-steroidal anti-inflammatory drugs (NSAIDs).
10. Subjects taking Phenytoin, calcium channel blockers drugs (CCBs) and/or cyclosporine, which might influence the pattern of tissue response.
11. Subjects treated with non-steroidal anti-inflammatory drugs (NSAIDs) within 14 days prior to entry into the study and throughout the study duration.
12. Presence of the following conditions: Type 1 diabetes, major recurrent aphtae, stomatitis, abscesses and related oral pathologies.
13. The presence of any medical or psychiatric condition that in the opinion of the investigator could affect the successful participation of the subject in the study.
14. Subject participates in any other clinical study 30 days prior to the start of the study and throughout the study duration.
15. Subject uses chlorhexidine oral rinses/ mouthwashes on a regular basis.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2009-08; Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Mean Probing Pocket Depth reduction | 8 weeks

SECONDARY OUTCOMES:
clinical attachment levels (CAL) and bleeding on probing (BOP) | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Periodontology, School of Graduate Dentistry, Rambam Health Care Center, Haifa, Israel